CLINICAL TRIAL: NCT02321553
Title: Biological Functions of Brown Rice on Metabolic Syndrome: A Randomized Cross-over Pilot Study
Brief Title: Effect of Brown Rice on the Risk Factors for Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Oliver Chen, Scientist I, Tufts University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 11066
Record Dates: First submitted 2014-12-10; First posted 2014-12-22 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; glucose; cholesterol; brown rice; inflammation; oxidative stress
MeSH Terms: conditions — Metabolic Syndrome; Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brown Rice (Experimental): Eat 100g of brown rice cake (3 packets) per day for 5 weeks
  Interventions: Other: Brown rice
- White Rice (Experimental): Eat 100g of white rice cake (3 packets) per day for 5 weeks
  Interventions: Other: White rice

INTERVENTIONS:
Other: Brown rice — brown rice cake
  Arms: Brown Rice
Other: White rice — white rice cake
  Arms: White Rice

SUMMARY:
The purpose of the study is to determine the effect of consumption of brown rice on the risk factors of metabolic syndrome (MetS) as compared to consumption of white rice. Brown and white rice will be provided in the form of rice cakes and 100g will be consumed per day for 5 weeks each. The investigators hypothesize that brown rice will have beneficial effects as it is rich in fiber and also phytochemicals.

DETAILED DESCRIPTION:
This is a 2-way cross-over, randomized, placebo controlled, pilot feasibility study to determine the effect of brown rice on the risk factors of metabolic syndrome (MetS). Eligible subjects (n = 9) with the MetS (>50 yr, post-menopausal women and men) will be randomized to receive either brown rice cakes (100 g/d) as treatment or white rice cake as placebo during each 5-wk intervention phase with a 2-wk washout between phases. Subjects will visit Tufts Medical Center for all study visits, at the end of baseline (first 2 week run in phase) and weeks 7, 9 and 14, which will include a 12 hour fasting blood draw. Two sets of three 24 hour dietary recalls will be conducted during the intervention phases. Fasting blood samples will be analyzed for 1) oxidative stress markers (vitamin E concentrations, total antioxidant capacity, and lipid peroxidation product), 2) blood lipid profiles and 3) metabolic risk factors such as plasma glucose, insulin, inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Men & postmenopausal women, aged >50 years
* BMI >30 kg/m2 and/or waist/hip ratio >0.9 for men, >0.85 for women
* plus any two of the following four MetS factors
* Fasting plasma TG: 150-400 mg/dL (1.7 - 4.52 mmol/L)
* Fasting plasma HDL cholesterol: <40 mg /dL (1.03 mmol/L) for men, <50 mg/dL (1.29 mmol/L) for women
* Blood pressure: SBP, 130-160 mmHg and/or DBP 85-95 mmHg
* Fasting plasma glucose: fasting blood glucose 100-125 mg/dL (5.55- 6.94 mmol/L) and no medication for blood glucose regulation and no use of insulin

Exclusion Criteria:

* Cigarette smoking and/or nicotine replacement use
* Individuals taking estrogen
* Use of blood glucose lowering medications or insulin
* Regular use (>2x/wk) of any stomach acid-lowering medications or laxatives
* Regular use (>2x/wk) of medication for inflammation
* Regular use of medication for hypercoagulation
* Cardiovascular (heart) disease
* Gastrointestinal disease
* Renal or chronic kidney disease
* Endocrine disease: including diabetes, untreated thyroid disease
* Rheumatoid arthritis
* Active treatment for any type of cancer, except basal cell carcinoma, within 1 year prior to study admission
* Systolic blood pressure >160 mmHg and/or diastolic blood pressure >95 mmHg
* Regular use of oral steroids except topical OTC steroids
* Regular daily intake of ≥2 alcoholic drinks
* Infrequent (<3/wk) or excessive (>3/d) number of regular bowel movements
* Illicit drug use
* Vegetarians
* No fish oil supplements (including cod liver oil) for one month prior to study admission
* No dietary supplements, including those containing any vitamins, minerals, herbs, plant concentrates (including garlic, gingko, St. John's wort) or homeopathic remedies, for one month prior to study admission
* On or planning a weight reducing regimen using a dietary approach of dietary supplements

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Glucoregulation (glucose, insulin and HbA1c) | Change from baseline after 5 week intervention phase

SECONDARY OUTCOMES:
Inflammatory markers (high sensitivity CRP, soluble intercellular adhesion molecule 1, serum amyloid A, vascular cell adhesion molecule 1) | Change from baseline after 5 week intervention phase
Lipid profile (Total cholesterol, HDL and Triglycerides) | Change from baseline after 5 week intervention phase
Oxidative stress markers - total antioxidant potential (TAP), total thiols, tocols, Ferric Reducing Antioxidant Power (FRAP), malondialdehyde (MDA), uric acid | Change from baseline after 5 week intervention phase

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Chen, Ph.D., Principal Investigator — Tufts University
Locations (1):
- Clinical and Translation Research Center, Tufts Medical Center, Boston, Massachusetts, United States